CLINICAL TRIAL: NCT00025623
Title: European Infant Neuroblastoma Study - Stage 4 With Bone, Lung, Pleura or CNS Involvement; MYCN Not Amplified
Brief Title: Combination Chemotherapy Followed by Surgery in Treating Infants With Newly Diagnosed Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Infant Neuroblastoma Study Group - 1999 (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068980; EURO-INF-NB-STUDY-1999-99.3; EU-20125C
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2002-12

CONDITIONS: Neuroblastoma
Keywords: disseminated neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Carboplatin; Cyclophosphamide; Doxorubicin; Etoposide; Vincristine

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: vincristine sulfate
Procedure: conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug, and giving them before surgery, may shrink the tumor so that it can be removed during surgery.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy followed by surgery in treating infants who have newly diagnosed neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Confirm that the management of infants with newly diagnosed stage IV neuroblastoma without MYCN amplification treated with etoposide and carboplatin and cyclophosphamide, doxorubicin, and vincristine followed by surgery does not require intensive high-dose chemotherapy consolidation.
* Determine whether deletion of chromosome 1p or diploidy/tetraploidy are prognostic factors in these patients.
* Determine whether there are other prognostic criteria that could be used in future therapeutic stratification of these patients.

OUTLINE: This is a multicenter study.

Patients receive VP-CARBO chemotherapy comprising etoposide IV over 2 hours and carboplatin IV over 1 hour on days 1-3. Treatment repeats every 21 days for 2 courses.

Patients without disease progression receive 2 additional courses of VP-CARBO chemotherapy. Patients with metastatic complete response (CR) undergo surgical resection of primary disease.

Patients with disease progression after 2 or 4 courses of VP-CARBO chemotherapy receive CADO chemotherapy comprising cyclophosphamide IV over 1 hour on days 1-5, doxorubicin IV over 6 hours on days 4 and 5, and vincristine IV on days 1 and 5. Treatment repeats every 21 days for 2 courses.

After 2 courses of CADO chemotherapy, patients with metastatic CR undergo surgical resection of primary disease. Patients with residual disease receive 2 additional courses of CADO chemotherapy. Patients with residual disease after 4 courses of CADO chemotherapy are removed from the study. Patients with metastatic CR after additional CADO chemotherapy undergo surgical resection of primary disease.

Patients are followed within 6 months and then annually for 5 years.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed stage IV neuroblastoma or ganglioneuroblastoma

  * Metastases to bone, CNS, or pleura/lung by x-ray or CT scan
* No MYCN amplification (i.e., fewer than 10 copies)

PATIENT CHARACTERISTICS:

Age:

* Under 12 months at diagnosis

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 1999-07; Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruno De Bernardi, MD, Study Chair — Istituto Giannina Gaslini
Locations (11):
- St. Anna Children's Hospital, Vienna, Austria
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Rigshospitalet, Copenhagen, Denmark
- Centre Hospitalier Regional de Purpan, Toulouse, France
- Istituto Giannina Gaslini, Genoa, Italy
- Rikshospitalet University Hospital, Oslo, Norway
- Instituto Portugues de Oncologia de Francisco Gentil - Centro Regional de Oncologia de Lisboa, S.A., Lisbon, Portugal
- Hospital Universitario LA FE, Valencia, Spain
- Ostra Sjukhuset, Gothenburg, Sweden
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland
- Bristol Royal Hospital for Children, Bristol, England, United Kingdom

REFERENCES:
- [Background] De Bernardi B, Gerrard M, Boni L, Rubie H, Canete A, Di Cataldo A, Castel V, Forjaz de Lacerda A, Ladenstein R, Ruud E, Brichard B, Couturier J, Ellershaw C, Munzer C, Bruzzi P, Michon J, Pearson AD. Excellent outcome with reduced treatment for infants with disseminated neuroblastoma without MYCN gene amplification. J Clin Oncol. 2009 Mar 1;27(7):1034-40. doi: 10.1200/JCO.2008.17.5877. Epub 2009 Jan 26. PMID 19171711